CLINICAL TRIAL: NCT04818684
Title: Practices of Accompaniment of the Relatives of Patients in the Agonic Phase by an Interdisciplinary Team
Acronym: PROPAGE2
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/60
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Practice Nurse's Scope
Keywords: Practices; accompaniment; interdisciplinary; relatives; agonic phase
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (7):
- Physician: at least 3 years of seniority in palliative care unit will be required, including 1 year in the participating palliative care unit.
  Interventions: Other: questionnaire
- Psychologists: at least 3 years of seniority in palliative care unit will be required, including 1 year in the participating palliative care unit.
  Interventions: Other: questionnaire
- Caregivers: at least 3 years of seniority in palliative care unit will be required, including 1 year in the participating palliative care unit.
  Interventions: Other: questionnaire
- Nurses: at least 3 years of seniority in palliative care unit will be required, including 1 year in the participating palliative care unit.
  Interventions: Other: questionnaire
- Social and Educational Assistants: at least 3 years of seniority in palliative care unit will be required, including 1 year in the participating palliative care unit.
  Interventions: Other: questionnaire
- Volunteers: at least 3 years of seniority in palliative care unit will be required, including 1 year in the participating palliative care unit. The representative participating in the study will preferably be the volunteer coordinator.
  Interventions: Other: questionnaire
- Relatives: Relative of a patient who died in the palliative care unit at least 6 months ago Person to trust or to prevent if not designated Relative understanding and speaking sufficient French Relative not a health professional
  Relative who visited the palliative care unit during the last 3 days of the patient's life and who met the care team:
  * Traceability of the arrival of the loved one in the last 2/3 days of the patient's hospitalization
  * Traceability of a meeting of the loved one with a member of the team over the last 3 days of his hospitalization or verification during telephone contact with the loved one after drawing lots Relative with an email address (to be verified during telephone contact with the loved one after drawing lots)
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — a questionnaire consisting of a list of support practices

SUMMARY:
The PROPAGE study program aims above all to improve the experience and satisfaction of family and friends regarding the support they receive during the dying person's agony phase.

DETAILED DESCRIPTION:
The objective of PROPAGE 2 is to establish a consensus on the practices for accompanying relatives during the agonic phase in the context of hospitalization in the palliative care unit by an interdisciplinary team.

ELIGIBILITY:
INCLUSION CRITERIA

1. PALLIATIVE CARE UNITS (USP) 35 palliative care unit will be drawn at random among the 164 French palliative care unit (www.sfap.org). In the event of refusal of participation, the drawing of lots will continue until 35 participating palliative care unit are obtained. The inclusion criteria for palliative care units were determined from the survey carried out in 2013 by the National End of Life Observatory on palliative care units in France. In order for there to be representativeness, the status of the palliative care unit will be taken into account from the national University Hospital (CHU) distribution, excluding CHU in the public sector, private non-profit sector, private for-profit sector. Thus, out of the 35 palliative care units: 7 will be within CHU, 16 will be outside CHU in the public sector, 7 will be in the private non-profit sector, and 5 in the private for-profit sector (criteria determined from the survey of the National End of Life Observatory in 2013) by ensuring that there are no more than 3 palliative care units in the same department (this in order to avoid that a geographical territory is over-represented, which would be liable to bias the results).

   In the event of refusal of a palliative care units or of inadequacy of the criteria, the drawing of lots will be continued until 35 participating USPs are obtained.

   Each team of these palliative care units must allow the participation of 7 experts: 1 for each group of experts, i.e. 5 socio-health professionals working in all the palliative care units (doctors, psychologists, nursing assistants, nurses, socio-educational assistant) as well as the coordinator of support volunteers and a relative by palliative care unit.
2. THE EXPERTS

6 volunteer experts who will participate in the panel of voters: a doctor (group 1), an IDE ( group 2), an AS (group 3), a psychologist (group 4), an ASE (group 5), a volunteer support coordinator (group 6) . A relative (group 7) will be done.

The inclusion criteria:

* For professionals, at least 3 years of seniority in palliative care unit will be required, including 1 year in the participating palliative care unit.
* For volunteers, at least 3 years of seniority in palliative care unit will be required, including 1 year in the participating palliative care unit. The representative participating in the study will preferably be the volunteer coordinator.
* For relatives Relative of a patient who died in the palliative care unit at least 6 months ago Person to trust or to prevent if not designated Relative understanding and speaking sufficient French Relative not a health professional

Relative who visited the palliative care unit during the last 3 days of the patient's life and who met the care team:

* Traceability of the arrival of the loved one in the last 2/3 days of the patient's hospitalization
* Traceability of a meeting of the loved one with a member of the team over the last 3 days of his hospitalization or verification during telephone contact with the loved one after drawing lots Relative with an email address (to be verified during telephone contact with the loved one after drawing lots)

NO-INCLUSION AND EXCLUSION CRITERIA

1. PALLIATIVE CARE UNITS Palliative care unit who could not be represented by the 7 experts required

   * Have participated in the PROPAGE 1 study
   * Have taken part in the questionnaire test.
2. THE EXPERTS Palliative care unit Experts: Anyone with less than 3 years of palliative care unit experience.

Relatives:

Relative of a patient who died in the palliative care unit less than 6 months ago Relative not understanding and not speaking French enough Relative being a health professional Relative who has not been to the palliative care unit in the last 3 days of the patient's life Relative who does not have an email address (to be checked during telephone contact with the loved one after drawing lots).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This includes people working in a palliative care unit as well as relatives who have known a patient in agony phase in a palliative care unit.
Sampling Method: Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Score of Likert-type scales (rated between 0 and 9), best match what each participant think about support practices for relatives of persons in the agony phase : from 1 (strongly disagree) to 9 (strongly agree). | Day 1
  It is based on a questionnaire made up of a list of support practices developed from the literature review and the list of practices identified through focus groups in the preliminary study PROPAGE 1. The responses are collected. on Likert-type scales reflecting the degree of agreement towards a proposition (rated between 0 and 9) and / or in the form of free comments.
Score of Likert-type scales (rated between 0 and 9), best match what each participant think about support practices for relatives of persons in the agony phase : from 1 (strongly disagree) to 9 (strongly agree). | Month 2
  It is based on a questionnaire made up of a list of support practices developed from the literature review and the list of practices identified through focus groups in the preliminary study PROPAGE 1. The responses are collected. on Likert-type scales reflecting the degree of agreement towards a proposition (rated between 0 and 9) and / or in the form of free comments.
Score of Likert-type scales (rated between 0 and 9), best match what each participant think about support practices for relatives of persons in the agony phase : from 1 (strongly disagree) to 9 (strongly agree). | Month 4
  It is based on a questionnaire made up of a list of support practices developed from the literature review and the list of practices identified through focus groups in the preliminary study PROPAGE 1. The responses are collected. on Likert-type scales reflecting the degree of agreement towards a proposition (rated between 0 and 9) and / or in the form of free comments.

CONTACTS AND LOCATIONS:
Overall Officials: Carole ROUMIGUIERE, Study Director — University Hospital, Bordeaux
Locations (1):
- Chu de Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No